CLINICAL TRIAL: NCT00394836
Title: A Single-arm, International, Multi-center Trial of HuMax-CD20, a Fully Human Monoclonal Anti-CD20 Antibody, in Patients With Follicular Lymphoma Who Are Refractory to Rituximab as Monotherapy or in Combination With Chemotherapy
Brief Title: HuMax-CD20 i(Ofatumumab) n Follicular Lymphoma (FL) Patients Refractory to Rituximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 111772; Hx-CD20-405 (Other: Genmab); 111772 (Other: GSK)
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2013-11

CONDITIONS: Lymphoma, Follicular
Keywords: ofatumumab; rituximab; NHL; CD20; refractory
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ofatumumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Ofatumumab — Eight weekly infusions of ofatumumab. The first infusion of 300mg ofatumunab
Drug: Ofatumumab — followed by 7 weekly infusions of 1000mg ofatumumab

SUMMARY:
A Single-Arm, International, Multi-Center Trial of HuMax-CD20 (Ofatumumab), a Fully Human Monoclonal Anti-CD20 Antibody, in Patients With Follicular Lymphoma Who Are Refractory to Rituximab as Monotherapy or in Combination With Chemotherapy

DETAILED DESCRIPTION:
Patients in the study will be randomized into two dose groups. Patients in each dose group will receive one infusion of 300 mg of HuMax-CD20 followed by 7 weekly infusions of either 500 or 1000 mg of HuMax-CD20. Disease status will be assessed every 3 months until month 24.

ELIGIBILITY:
Inclusion Criteria

* Patient with follicular lymphoma grade 1 - 2
* Refractory to rituximab given as monotherapy or in combination with any chemotherapy or to rituximab given as maintenance treatment following R-chemo, defined as:
* failure to achieve at least PR to rituximab given as monotherapy or in combination with any chemotherapy; or,
* disease progression while on rituximab (either given as monotherapy or in combination with any chemotherapy or during rituximab maintenance treatment following R-chemo); or,
* disease progression in responders within 6 months of the last dose of rituximab (either given as monotherapy or in combination with any chemotherapy or after rituximab maintenance treatment schedule following R-chemo)
* Tumor verified to be CD20+ positive from excisional lymph node biopsy
* CT scan in screening phase (based on local evaluation) showing:
* 2 or more clearly demarcated lesions with a largest diameter ≥ 1.5 cm, or
* 1 clearly demarcated lesion with a largest diameter ≥ 2,0 cm
* ECOG Performance Status of 0, 1, or 2
* Age ≥ 18 years
* Following receipt of verbal and written information about the study, the patient must provide signed informed consent before any study related activity is carried out

Exclusion Criteria

* Previous autologous stem cell transplantation within 6 months
* Previous allogeneic stem cell transplantation
* More than 1 previous radio immunotherapy regimen
* Received radio immunotherapy within 3 months
* Received any Anti-cancer treatment within 4 weeks
* Received monoclonal antibodies, other than rituximab within 3 months
* Patients previously treated with anti-CD20 monoclonal antibodies, other than rituximab
* Life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2007-05; Primary Completion 2009-04 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Southampton, United Kingdom

REFERENCES:
- [Background] Czuczman MS, Fayad L, Delwail V, Cartron G, Jacobsen E, Kuliczkowski K, Link BK, Pinter-Brown L, Radford J, Hellmann A, Gallop-Evans E, DiRienzo CG, Goldstein N, Gupta I, Jewell RC, Lin TS, Lisby S, Schultz M, Russell CA, Hagenbeek A; 405 Study Investigators. Ofatumumab monotherapy in rituximab-refractory follicular lymphoma: results from a multicenter study. Blood. 2012 Apr 19;119(16):3698-704. doi: 10.1182/blood-2011-09-378323. Epub 2012 Mar 2. PMID 22389254

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to one of two ofatumumab dose arms. Disease progression and treatment refusal resulted in some participants entering early follow up after early withdrawal from study treatment. They are being followed for overall survival.
Groups:
- Ofatumumab 500 mg: Ofatumumab intravenous (iv) infusion initiated at 300 milligrams (mg), followed by an infusion of 500 mg administered once weekly for 7 infusions. In the extended follow-up phase of the study, participants were followed only for survival status for up to 5 years and new follicular lymphoma (FL) treatment. Time to the next FL treatment analysis included participants which received new FL treatment during extended follow-up.
- Ofatumumab 1000 mg: Ofatumumab iv infusion initiated at 300 mg, followed by an infusion of 1000 mg administered once weekly for 7 infusions. In the extended follow-up phase of the study, participants were followed only for survival status for up to 5 years and new Follicular lymphoma (FL) treatment. Time to the next FL treatment analysis included participants which received new FL treatment during extended follow-up.
Period: Teatment or Follow-up Phase
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Started | 30 | 86
Early Follow-up Entry | 4 (Did not complete treatment.) | 8 (Did not complete treatment.)
Completed | 2 | 8
Not Completed | 28 | 78
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Disease Progression | 27 | 60
Not completed — Patient Refusal | 1 | 2
Not completed — Death | 0 | 1
Not completed — Patient refuses to continue with CT scan | 0 | 1
Not completed — Started alternative treatment | 0 | 6
Not completed — Suspicion of cholangiocarcinoma | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Patient progressed, return to Pakistan | 0 | 1
Not completed — Non compliance | 0 | 1
Period: Extended Follow-up Phase (2-5 Years)
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Started | 20 (Not all participants went into extended follow up per protocol.) | 58 (Not all participants went into extended follow up per protocol.)
Completed | 0 | 5
Not Completed | 20 | 53
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 0 | 1
Not completed — Alternative treatment | 13 | 41
Not completed — Medical Reasons | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Ofatumumab 500 mg: Ofatumumab intravenous (iv) infusion initiated at 300 milligrams (mg), followed by an infusion of 500 mg administered once weekly for 7 infusions
- Ofatumumab 1000 mg: Ofatumumab iv infusion initiated at 300 mg, followed by an infusion of 1000 mg administered once weekly for 7 infusions
- Total: Total of all reporting groups
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg | Total
Number analyzed (Participants) | 30 | 86 | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (10.1) | 59.7 (11.1) | 59.9 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 43 | 54
  Male | 19 | 43 | 62
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 4 | 5
  Black or African American | 0 | 1 | 1
  Hispanic or Latino | 0 | 3 | 3
  White | 28 | 78 | 106
  Reunion Island Native | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response (OR)
Description: OR was assessed by an Independent endpoints Review Committee (IRC) according to the standardized response criteria for Non-Hodgkin's lymphoma. Participants with Complete Response (CR; complete disappearance of all detectable disease), Complete Response unconfirmed (CRu; any residual lymph node/nodal mass >1.5 centimeters [cm] in its longest transverse diameter that regressed >75% compared to baseline), or Partial Response (PR; >=50% decrease in the sum of the product of diameters of indicator lesions) were defined as responders for OR.
Time Frame: Start of treatment (Day 1 of Week 0) until 3 months after start of last infusion (up to Week 32)
Population: Full Analysis Set (FAS): all participants who were exposed to study drug irrespective of their compliance to the planned course of treatment
Measure: Number; unit: participants
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 30 | 86
participants
  CR | 0 | 1
  CRu | 2 | 0
  PR | 2 | 8
Statistical Analysis 1: Comparison: Ofatumumab 500 mg; Test type: Superiority or Other; percentage of responders = 13, 95% CI 2-sided [4 to 31] — Response rate is calculated as the number of responses divided by the number of participants treated * 100
Statistical Analysis 2: Comparison: Ofatumumab 1000 mg; Test type: Superiority or Other; percentage of responders = 10, 95% CI 2-sided [5 to 19]

2. Primary Outcome: Number of Participants Classified as Responders and Non-responders for Objective Response (OR)
Description: Based on OR over a 6-month period from start of treatment, participants were classified as responders/non-responders as follows: participants with CR, CRu, or PR were classified as responders, whereas participants with Stable Disease (SD; achieving less than PR but not consistent with PD), Progressive Disease (PD; 50% increase from nadir in the products of the greatest perpendicular diameters of any previously identified node or appearance of any new node >1 cm), or Not Evaluable (NE) participants were classified as non-responders.
Time Frame: 6-month period from the start of treatment. There was a median time of response at Month 5.5 (participants were followed for up to 24 months).
Population: FAS
Measure: Number; unit: participants
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 30 | 86
participants
  Responders with CR | 0 | 1
  Responders with CRu | 2 | 0
  Responders with PR | 2 | 8
  Non-responders with SD | 9 | 43
  Non-responders with PD | 14 | 26
  Non-responders with NE | 3 | 8

3. Secondary Outcome: Duration of Response
Description: The duration of response is defined as the time from the initial response (the first visit at which response was observed) to progression or death. For participants who were lost to follow-up, duration of response was censored at the date of the last attended visit at which the endpoint was assessed. The Kaplan-Meier method was used to estimate duration of response.
Time Frame: From start of treatment (Week 0) until Month 24
Population: FAS. Only those participants classified as responders were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 4 | 9
months | 6.0 [2.9 to 6.2] | 6.0 [2.8 to 12.3]

4. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) is defined as the time from randomization until the first radiologically or clinically documented evidence of progression or death due to any cause, if sooner. For participants who were lost to follow-up, PFS was censored at the date of the last attended visit at which the endpoint was assessed. The Kaplan-Meier method was used to estimate PFS.
Time Frame: From start of treatment (Week 0) until Month 24
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 30 | 86
Months | 3.2 [2.9 to 9.2] | 6.0 [4.4 to 9.0]

5. Secondary Outcome: Time to Next Follicular Lymphoma (FL) Therapy
Description: Time to next FL (anti-lymphoma) therapy is defined as the time from randomization until the time of first administration of the next anti-lymphoma therapy other than ofatumumab. For participants who were lost to follow-up, the time was censored at the date of the last attended visit at which the endpoint was assessed.
Time Frame: From start of treatment (Week 0) until Month 24
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 30 | 86
Months | 4.2 [3.8 to 8.6] | 7.0 [5.5 to 9.9]

6. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization until death. For participants who are lost to follow-up, overall survival will be censored at the date of the last attended visit at which the endpoint was assessed.
Time Frame: First dose (Week 0) until 5 years
Population: FAS. As of the time of data cut-off, data for Overall Survival was not estimable because too few deaths have occurred at the time of study completion.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 30 | 86
Months | NA [NA to NA] — Overall survival was not estimable due to too few deaths.; therefore the median and CI cannot be calculated. | NA [NA to NA] — Overall survival was not estimable due to too few deaths.; therefore the median and CI cannot be calculated.

7. Secondary Outcome: Percent Change From Screening (Visit 1) in Tumor Size as Assessed by Radiologist 1 (R1) and Radiologist 2 (R2) at Months 3, 6, 9, 12, 18, and 24
Description: Tumor size was measured by computed tomography (CT) scan and was computed as the sum of product of diameters (SPD) for the indicator lesions. CT scans with contrast of the neck, thorax, abdomen, and pelvis were performed at Screening and during the follow-up period (Month 3, 6, 9, 12, 18, and 24). The change in tumor size from Screening (Visit 1) was presented per Radiologist 1 (R1) and Radiologist 2 (R2). Percent change from Screening (Visit 1, Week -2) = (value at Visits 11, 12, 13, 14, 16, and 18 minus the value at Visit 1 divided by the value at Visit 1) * 100.
Time Frame: Visits 1 (Week -2), 11 (Month 3), 12 (Month 6), 13 (Month 9), 14 (Month 12), 16 (Month 18), and 18 (Month 24)
Population: FAS. Data were provided for the number of participants attending each visit. Participants withdrawn during the study were not analyzed.
Measure: Median (Full Range); unit: percent change in tumor size
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 15 | 47
percent change in tumor size
  Visit 11 (Month 3), R1, n=14, 47 | 5.50 [-85.00 to 52.00] | -7.20 [-66.00 to 69.00]
  Visit 11 (Month 3), R2, n=15, 47 | -2.10 [-84.00 to 27.00] | -8.10 [-82.00 to 56.00]
  Visit 12 (Month 6), R1, n=7, 34 | -20.30 [-90.00 to 13.00] | -16.10 [-91.00 to 123.00]
  Visit 12 (Month 6), R2, n=7, 33 | -39.90 [-86.00 to 29.00] | -29.80 [-83.00 to 61.00]
  Visit 13 (Month 9), R1, n=6, 25 | -28.90 [-85.00 to 30.00] | -22.60 [-88.00 to 138.00]
  Visit 13 (Month 9), R2, n=6, 26 | -48.30 [-84.00 to 34.00] | -39.80 [-85.00 to 91.00]
  Visit 14 (Month 12), R1, n=4, 17 | 5.50 [-69.00 to 74.00] | -16.00 [-73.00 to 42.00]
  Visit 14 (Month 12), R2, n=4, 18 | -14.70 [-83.00 to 63.00] | -44.60 [-91.00 to 62.00]
  Visit 16 (Month 18), R1, n=3, 12 | 31.10 [-81.00 to 202.00] | -18.30 [-49.00 to 45.00]
  Visit 16 (Month 18), R2, n=3, 12 | 22.90 [-87.00 to 52.00] | -28.70 [-91.00 to 50.00]
  Visit 18 (Month 24), R1, n=2, 8 | -4.80 [-85.00 to 75.00] | -20.10 [-64.00 to 4.00]
  Visit 18 (Month 24), R2, n=2, 8 | -14.40 [-88.00 to 59.00] | -36.50 [-92.00 to 35.00]

8. Secondary Outcome: Percent Change From Baseline (Visit 2) in CD19+ and CD20+ Cells in Peripheral Blood at Visits 11 and 12
Description: CD19 and CD20 are proteins found on the cell surface of B cells, and they can be detected in peripheral blood by flow cytometry. Flow cytometry of peripheral blood was performed for immediate analysis of cells with cluster of differentiation 19 (CD19+) and CD20+. The analysis will be done until a value is reached that is in the normal range. Percent change from Baseline (Visit 2) = (value at Visits 11 and 12 minus the value at Visit 2 divided by the value at Visit 2) * 100.
Time Frame: Visits 2 (Baseline), 11 (Month 3), and 12 (Month 6)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: percent change in cells
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 15 | 45
percent change in cells
  Visit 11 (Month 3), CD19+, n=15, 42 | -100.00 [-100.00 to 0.00] | -80.1 [-100.00 to 566.00]
  Visit 11 (Month 3), CD20+, n=15, 45 | -100.00 [-100.00 to 0.00] | -100.00 [-100.00 to 43.00]
  Visit 12 (Month 6), CD19+, n=8, 32 | -48.80 [-100.00 to 129.00] | -19.00 [-100.00 to 838.00]
  Visit 12 (Month 6), CD20+, n=8, 34 | -48.20 [-100.00 to 129.00] | -19.00 [-100.00 to 18.00]

9. Secondary Outcome: Number of Participants With Conversion and no Conversion of BCL2 Positive to BCL2 Negative in Peripheral Blood
Description: B-cell lymphoma 2 (BCL2) is the second member of a range of proteins initially described in chromosomal translocations involving chromosomes 14 and 18 in follicular lymphomas. BCL2 mitochondrial ribonucleic acid (mRNA) was measured by polymerase chain reaction (PCR) from peripheral blood. Participants who had no post-screening data were categorized as "Missing."
Time Frame: Screening (Visit 1) until Month 24 (Visit 18)
Population: FAS. Only those participants who were BCL2 positive at Screening were analyzed.
Measure: Number; unit: participants
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 11 | 31
participants
  Participants converted from positive to negative | 2 | 6
  Participants not converted | 6 | 15
  Missing | 3 | 10

10. Secondary Outcome: Number of Participants Who Experienced Any Adverse Event From First Treatment (Visit 2) to Visit 18 (Month 24)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. A list of AEs experienced in the study at a frequency threshold of 5% can be found in the AE section.
Time Frame: From first treatment (Visit 2) until Visit 18 (Month 24)
Population: FAS
Measure: Number; unit: participants
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 30 | 86
participants | 30 | 79

11. Secondary Outcome: Number of Participants With Positive Human Anti-human Antibodies (HAHA) at Visits 1, 12, 13, and 14
Description: HAHA are indicators of immunogenicity to ofatumumab. Blood samples were withdrawn from participants at Visits 1, 12, 13, and 18 for analysis of HAHA. Analysis of HAHA was done in batches.
Time Frame: Visits 1 (Screening), 12 (Month 6), 13 (Month 9), and 18 (Month 24)
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 30 | 85
participants
  Visit 1 (Week -2), n=30, 85 | 0 | 0
  Visit 12 (Month 6), n=8, 33 | 0 | 0
  Visit 13 (Month 9), n=7, 24 | 0 | 0
  Visit 14 (Month 12), n=3, 11 | 0 | 0

12. Secondary Outcome: Complement (CH50) Levels at Visit 1 and at the End of Infusion at Visit 2
Description: Blood samples were drawn from participants at Visits 1 and 2 for analysis of complement (CH50) levels. Analysis of CH50 was done in batches, and CH50 levels were measured two hours after the end of study medication infusion. Percent change from Screening (Visit 1, Week -2) = (value at Visit 2 minus the value at Visit 1 divided by the value at Visit 1) * 100.
Time Frame: Visits 1 (Week -2) and 2 (Week 0)
Population: as for outcome 7
Measure: Median (Full Range); unit: Units per milliliter (U/mL)
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 30 | 85
Units per milliliter (U/mL)
  Visit 1 (Week -2), n=30, 85 | 57.00 [10.00 to 79.00] | 54.00 [10.00 to 99.00]
  Visit 2 (Week 0), n=30, 84 | 49.00 [10.00 to 76.00] | 49.50 [10.00 to 92.00]

13. Secondary Outcome: Number of Participants Classified as Responders for Fragment C Receptor (FcR) Polymorphism (Poly.)
Description: FcR poly. affect the affinity with which FcRs interact with immunoglobulin molecules and are prognostic factors that are indicative of altered responsiveness to treatment and/or survival. A blood sample was drawn at Visit 1 for analysis (done in batches of several samples) of FcR poly. (Fcgamma RIIIa Valine/Phenylalanine genotypes [TT=thymidine/thymidine, TG=thymidine/guanine, GG=guanine/guanine] and Fcgamma RIIa Arginine/Histidine genotypes [AA=adenine/adenine, AG=adenine/guanine, GG=guanine/guanine]). Responders must have met the criteria for CR, CRu, or PR at either Month 3 or Month 6. Fc receptor polymorphisms and C1qA-276 results are not included in this results summary.
Time Frame: From first treatment (Visit 2) until Visit 12 (Month 6)
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 11 | 37
participants
  Fc Gamma IIa Genotype = AA, n=4, 9 | NA — Proper informed consent was not obtained; therefore, we cannot use these data. | NA — Proper informed consent was not obtained; therefore, we cannot use these data.
  Fc Gamma IIa Genotype = AG, n=11, 37 | NA — Proper informed consent was not obtained; therefore, we cannot use these data. | NA — Proper informed consent was not obtained; therefore, we cannot use these data.
  Fc Gamma IIa Genotype = GG, n=3, 12 | NA — Proper informed consent was not obtained; therefore, we cannot use these data. | NA — Proper informed consent was not obtained; therefore, we cannot use these data.
  Fc Gamma IIIa Genotype = TT, n=5, 31 | NA — Proper informed consent was not obtained; therefore, we cannot use these data. | NA — Proper informed consent was not obtained; therefore, we cannot use these data.
  Fc Gamma IIIa Genotype = TG, n=11, 23 | NA — Proper informed consent was not obtained; therefore, we cannot use these data. | NA — Proper informed consent was not obtained; therefore, we cannot use these data.
  Fc Gamma IIIa Genotype = GG, n=2, 4 | NA — Proper informed consent was not obtained; therefore, we cannot use these data. | NA — Proper informed consent was not obtained; therefore, we cannot use these data.

14. Secondary Outcome: Ctrough and Cmax at the Eighth Infusion (Visit 9, Week 7)
Description: Cmax is defined as the maximum concentration of drug in plasma samples. Ctrough is defined as the trough plasma concentration (measured concentration at the end of a dosing interval [taken directly before the start of the next infusion]).
Time Frame: Visit 9 (Week 7; up to 10 months after dose)
Population: FAS. Data were provided for the number of participants who had a value. Cmax was not reported for one participant due to missing data. Participants withdrawn during the study were not analyzed. Interim results; data as of 28 April 2009.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams per liter (mg/L)
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 24 | 78
Milligrams per liter (mg/L)
  Ctrough, n=24, 78 | 183 (3.40) | 447 (1.31)
  Cmax, n=23, 78 | 479 (0.40) | 879 (0.45)

15. Secondary Outcome: AUC(0-inf) and AUC(0-168) After the Eighth Infusion (Visit 9, Week 7)
Description: AUC is defined as the area under the ofatumumab concentration-time curve as a measure of drug exposure. AUC(0-168) is AUC from the start of infusion to 168 hours after the start of the infusion; AUC(0-inf) is AUC from the start of infusion extrapolated to infinity.
Time Frame: Visit 9 (Week 7; up to 10 months after dose)
Population: FAS. Data were provided for the number of participants for whom the parameter could be calculated. Participants withdrawn during the study were not analyzed. Interim results; data as of 28 April 2009.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams * hour per liter (mg.h/L)
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 19 | 75
Milligrams * hour per liter (mg.h/L)
  AUC(0-inf), n=12, 55 | 327715 (1.03) | 566717 (1.07)
  AUC(0-168), n=19, 75 | 71513 (0.40) | 113622 (0.65)

16. Secondary Outcome: t1/2 After the Eighth Infusion (Visit 9, Week 7)
Description: t1/2 is defined as terminal half-life, which is the time required for the amount of the drug in the body to decrease by half.
Time Frame: Visit 9 (Week 7; up to 10 months after dose)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 12 | 55
hours | 444 (0.76) | 443 (0.64)

17. Secondary Outcome: CL After the Eighth Infusion (Visit 9, Week 7)
Description: CL is the clearance of drug from plasma, which is defined as the volume of plasma from which drug is removed per unit time.
Time Frame: Visit 9 (Week 7; up to 10 months after dose)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliters per hour (mL/h)
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 18 | 75
Milliliters per hour (mL/h) | 7.0 (0.41) | 8.8 (0.65)

18. Secondary Outcome: Vss After the Eighth Infusion (Visit 9, Week 7)
Description: Vss is the volume of distribution at steady state of ofatumumab.
Time Frame: Visit 9 (Week 7; to up 10 months after dose)
Population: FAS. Data were provided for the number of participants for whom the parameter could be calculated. Participants withdrawn during the study were not analyzed. Interim results; data of 28 April 2009.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg
Number analyzed (Participants) | 11 | 55
mL | 4414 (0.48) | 5408 (0.34)

ADVERSE EVENTS:
Description: During the Extended Follow-up Phase, from 2 years to 5 years after first treatment, only serious adverse events (SAEs) were collected; no non-serious AEs were collected during this period.
Groups:
- Ofatumumab 500 mg: Extended Follow-up Phase: Ofatumumab intravenous (iv) infusion initiated at 300 milligrams (mg), followed by an infusion of 500 mg administered once weekly for 7 infusions. In the extended follow-up phase of the study, participants were followed only for survival status for up to 5 years and new follicular lymphoma (FL) treatment. Time to the next FL treatment analysis included participants which received new FL treatment during extended follow-up.
- Ofatumumab 1000 mg: Extended Follow-up Phase: Ofatumumab iv infusion initiated at 300 mg, followed by an infusion of 1000 mg administered once weekly for 7 infusions. In the extended follow-up phase of the study, participants were followed only for survival status for up to 5 years and new Follicular lymphoma (FL) treatment. Time to the next FL treatment analysis included participants which received new FL treatment during extended follow-up.
Arm/Group | Ofatumumab 500 mg | Ofatumumab 1000 mg | Ofatumumab 500 mg: Extended Follow-up Phase | Ofatumumab 1000 mg: Extended Follow-up Phase
Serious Adverse Events (participants affected / at risk) | 6/30 | 25/86 | 2/30 | 6/86
Other Adverse Events (participants affected / at risk) | 30/30 | 79/86 | 0/30 | 0/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab 500 mg (N=30) | Ofatumumab 1000 mg (N=86) | Ofatumumab 500 mg: Extended Follow-up Phase (N=30) | Ofatumumab 1000 mg: Extended Follow-up Phase (N=86)
Disease progression (General disorders) | 2 | 4 | 1 | 3
Generalised oedema (General disorders) | 0 | 1 | 0 | 0
Hypothermia (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 5 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 2 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Neutropenic infection (Infections and infestations) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0
Progressive Multifocal Leukoencephalopathy (Infections and infestations) | 0 | 0 | 0 | 1
Blindness (Eye disorders) | 0 | 0 | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab 500 mg (N=30) | Ofatumumab 1000 mg (N=86) | Ofatumumab 500 mg: Extended Follow-up Phase (N=30) | Ofatumumab 1000 mg: Extended Follow-up Phase (N=86)
Fatigue (General disorders) | 4 | 13 | 0 | 0
Asthenia (General disorders) | 2 | 11 | 0 | 0
Oedema peripheral (General disorders) | 6 | 7 | 0 | 0
Pyrexia (General disorders) | 2 | 11 | 0 | 0
Disease progression (General disorders) | 2 | 4 | 0 | 0
Chest discomfort (General disorders) | 2 | 2 | 0 | 0
Chest pain (General disorders) | 2 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 14 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 12 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 10 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 5 | 4 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 6 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 2 | 0 | 0
Headache (Nervous system disorders) | 4 | 7 | 0 | 0
Paraesthesia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 10 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 8 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 5 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 7 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 6 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 6 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 4 | 0 | 0
Hypotension (Vascular disorders) | 1 | 5 | 0 | 0
Flushing (Vascular disorders) | 2 | 3 | 0 | 0
Hypersensitivity (Immune system disorders) | 3 | 6 | 0 | 0
Hematuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Chills (General disorders) | 1 | 5 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.